CLINICAL TRIAL: NCT02857972
Title: Proof of Concept Study of Wondaleaf® As an Alternative to Menstrual Hygiene Product for Night Use Among Menstruating Women
Brief Title: Proof Of Concept Menstrual Hygiene Product-Wondaleaf®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Twin Catalyst Sdn. Bhd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRR-16-239-29465
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Other Menstruation Disorders
Keywords: Menstruation, Female Barrier, Sanitary pads

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wondaleaf® (Experimental): This is a single arm clinical trial, all female subjects will be recruited to the arm using investigational device only.
  Interventions: Device: Wondaleaf®

INTERVENTIONS:
Device: Wondaleaf® — Use of Wondaleaf® during menstruation every night in one menstrual cycle.
  Other Names: Female Barrier Film

SUMMARY:
General objective:

To assess the preference and performance in terms of satisfaction and acceptability as well as safety profile of a novel innovative design of menstrual hygiene device (Wondaleaf®) during the night for menstruating women by comparing it to prior experience of the usual hygienic product for menstrual control, i.e. sanitary pads.

Specific objectives:

* To determine the preference of participants between Wondaleaf® and usual sanitary pads as a night use menstrual hygiene product.
* To determine the satisfaction of participants towards Wondaleaf® and usual sanitary pads as a night use menstrual hygiene product.
* To determine the acceptability of participants towards Wondaleaf® as a night use menstrual hygiene product.
* To determine the safety profile of the Wondaleaf®.

DETAILED DESCRIPTION:
This is a proof of concept study to assess preference, satisfaction and acceptability of Wondaleaf® versus prior experience of sanitary pads for night use among menstruating women. Community sampling will be done and 30 women within ages of 18 to 45 years old with regular menstrual cycles will be recruited. Potential participants will be screened based on the inclusion and exclusion criteria.

During the Visit 1 after recruitment, participants will have to complete the Baseline Questionnaire (Refer to Appendix):

Table 1 - Socio-demographic: age, race, education level, marital and personal / family income status.

Table 2 - Usual menstrual characteristics for the past 1 year: age of menarche; most frequent length of menstrual cycle (days); most frequent duration of each menstrual bleeding (days); number of days with heavy bleeding; the usual (i.e. commonest types) of sanitary pads used at night (panty liner, ultra-thin, regular, maxi / super or night use); estimated number of times hygiene product changed at night with heavy bleeding; estimated number of times hygiene product changed at night with average menstrual flow and current menstrual problems if any.

Table 3 - satisfaction of usual sanitary pads usage: product comfort; cleanliness; capacity; convenience; appearance and quality.

Participants will receive instructions and demonstrations regarding the investigational device usage. Any update on the device will be informed by research officers through phone call. Each women subject is required to use the investigational device given for the subsequent menstrual cycle at night and record the day of the menstrual flow starts and ends with the frequency of the device changed for each night in the Wondaleaf® Menstrual Diary. The test materials that are used shall be discarded appropriately in the usual manner at home.

A Home-based Questionnaire on the safety of the investigational device has to be completed by the participants at home within 24 hours of the last usage of Wondaleaf®.

Satisfaction, acceptability and preference questionaire will be given at Visit 2 at the end of menstrual cycle within 7 days following the last use of Wondaleaf®. Any unused investigational devices will be returned for counting purposes.

A final follow up by a phone call to each subject will be performed to enquire their general well-being after 3 months (+/- 7 days) of last Wondaleaf® usage.

If the women were confirmed pregnant during study duration, the subject will be withdrawn from the study and referred for antenatal care of their choice. If any adverse event arises, subject will be advised to stop using the investigational device and will be referred for medical care in the Hospital by relevant specialist.

ELIGIBILITY:
Inclusion Criteria:

1. Women within ages of 18 to 45 years old with good health and regular menstrual cycles with last menstrual cycle occurred within 5 weeks of enrolment; subjects can be rescreened after completion of menstrual cycle
2. Women who use sanitary pads as their only menstrual hygiene product.
3. Women who agree to use only the study menstrual hygiene device and not sanitary pads or other menstrual hygiene products for menstruation during the night time of study duration.
4. Women who are able to understand instructions for correct use of study menstrual hygiene product (i.e. the investigational device).
5. Literate women who can complete the study questionnaire on their own in a language of their choice which are English, Malay and Chinese; and attending all study visits.

Exclusion Criteria:

1. Known history of vaginal or uterine infection(s), and/or urinary tract infections; these subjects can be rescreened after 14 days after successful treatment.
2. Ongoing or past history of sexually transmitted disease, pelvic inflammatory disease, and/or injuries to the pelvis requiring surgical intervention and/or pelvic floor physiotherapy.
3. Female subject who is pregnant (established by urinary pregnancy test).
4. Sensitivity or allergy to polyurethane and acrylic adhesive hypoallergenic.
5. Staff who work directly under the investigators and/or employed directly by the device manufacturers, sponsor and study team.
6. Moving outside Sibu area during study period and have difficulty to return for Visit 2.
7. Female subjects who have menopause (absence of menstruation for more than 6 months in female) or any other circumstances that cause secondary amenorrhea (absence of menstruation for more than 6 months in a normal female of reproductive age that is not due to pregnancy) such as side effect from hormonal contraceptive.
8. Use any medications or preparation applied topically to the perineum or intravaginally to the genitalia but subjects can be rescreened 14 days after the recovery if the application is for acute illness.
9. Use of any medications which known to influence menstruation or study results for any reasons within 14 days, 30 days before Visit 1 and during the intended study duration.
10. Subject participating in another clinical study involving menstrual hygiene device.
11. Acute disease at the time of enrolment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. Fever is defined as axillary / tympanic / rectal temperature ≥ 38°C. Subjects can be rescreened 14 days after the recovery;
12. Blood dyscrasias, bleeding disorder, leukaemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems;
13. Presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, hepatic, immunologic, hematological, endocrine, or nervous system(s) or psychiatric disease or other conditions that may interfere with the health conditions (such as in case the women subject become pregnant), or would place the subjects at increased risk, as determined by the investigator(s).

Significant is defined as any disease/condition that, in the opinion of the researcher, would put the subject's safety at risk through study participation, or which would confound the interpretation of the study results if the disease/condition exacerbated during the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Preference | every night for one cycle of menstruation, an average of 5 days
  Wondaleaf® usage during the night is better; same or worse as compared to usual sanitary pad usage during menstruation.

SECONDARY OUTCOMES:
Satisfaction | every night for one cycle of menstruation, an average of 5 days
  Wondaleaf® 's comfort, cleanliness, capacity, convenience, appearance and quality on a 10-point sliding scale scoring with "1" for very poor to "5" being average up to "10" for very good as compare to experience of usual sanitary pads.
Acceptability | every night for one cycle of menstruation, an average of 5 days
  Likert scale scoring with scores of "1" being not likely to"5" being very likely whether subjects will continue, recommend or buy the device in the future.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | every night for one cycle of menstruation till 3 months after last usage of investigational device
  Monitoring adverse event locally at the perineum, vaginal infection or discharge and/or urinary tract infections and recording all adverse events, serious adverse events, adverse device events and serious adverse device events throughout the therapy session and immediately following therapy: allergy to Wondaleaf® and any systemic reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Teck Hock Toh, Principal Investigator — Clinical Research Centre, Sibu Hospital, Sarawak State Health Department, Ministry of Health Malaysia; Vivian Wee Yen Tan, Principal Investigator — Clinical Research Centre, Sibu Hospital, Sarawak State Health Department, Ministry of Health Malaysia
Locations (1):
- Sibu Hospital, Sibu, Sarawak, Malaysia